CLINICAL TRIAL: NCT02697097
Title: Muscle Strength in Femoroacetabular Impingement: A Comparative Study of Patients With FAI Versus Normal Controls
Brief Title: Hip Muscle Strength in FAI Versus Normal Controls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Vikas Khanduja MA FRCS (Orth), Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: AddenbrookesH
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Femoro-acetabular Impingement
Keywords: Hip Muscle Strength; FAI
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Arm Group: Participants aged 18-30, Male and Female (10 participants each). Control group must have normal range of movement and no evidence of femoro-acetabular impingement (FAI) on clinical examination (negative impingement test, no symptoms). Other exclusions for Control Group include previous surgery to hip joint/s, history of arthritis, family history of FAI, patients who have had symptoms of hip pain in the preceding 1 year or may have other conditions which may affect the hip joint or hip muscle strength including neurological conditions or muscular dystrophy.
- FAI Arm Comparison Group: Participants aged 18-30, Male and Female (10 participants each). Participants with femoro-acetabular impingement as diagnosed clinically and on radiological imaging for the comparison group (MRI).

SUMMARY:
Hip Muscle Strength in femoro-acetabular impingement participants versus normal controls.

To investigate the hip muscle strength in a normal control group and compare this to patients who have a diagnosis of femoro-acetabular impingement (diagnosed clinically and with confirmed radiological features).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females.
* Aged 18-30.
* Control group - Normal range of movement and no evidence of femoro-acetabular impingement on clinical examination (negative impingement test, no symptoms).
* Participants with femoro-acetabular impingement as diagnosed clinically and on radiological imaging for the comparison group (MRI).

Exclusion Criteria:

* Patients under the age of 18.
* Patients over the age of 30.
* Control group - evidence of underlying pathology affecting the hip, abnormal range of motion, evidence of femoro-acetabular impingement on clinical examination.
* Previous surgery of the hip joints.
* Medical history of arthritis (including rheumatoid and reactive).
* Family history of femoro-acetabular impingement (control arm participants).
* Patients who are currently experiencing or have experienced hip pain in the previous 1 year (control arm).
* Other conditions (e.g. neurological, muscular dystrophy etc) which may affect hip muscle strength.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control Arm Group - Medical Students who fit the inclusion criteria and are between ages of 18-30.
  FAI Comparison Group - Participants will be recruited from Young Adult Hip Clinic, meeting the defined inclusion criteria and also being between the ages of 18-30.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength on Dynamometer | 3 months

SECONDARY OUTCOMES:
Kinematics of the Hip - Range of Movement | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Khanduja, MA, FRCS (Orth), Principal Investigator — Consultant Trauma and Orthopaedic Surgeon - Principal Investigator
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No